CLINICAL TRIAL: NCT02042573
Title: TMSFOS: Preliminary Study to Investigate the Effect of rTMS and SSRI Antidepressants on Leukocyte Expression of the C-FOS and DUSP1 Genes in Patients Treated for Depression
Brief Title: Preliminary Study to Investigate the Effect of rTMS and SSRI Antidepressants on Leukocyte Expression of the C-FOS and DUSP1 Genes in Patients Treated for Depression
Acronym: TMSFOS
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study population is no longer accessible to the investigating team.
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: TROJAK APJ 2012
Record Dates: First submitted 2014-01-17; First posted 2014-01-23 (Estimated); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Selective Serotonin Reuptake Inhibitors

ARMS (3):
- Depressive patients treated with rTMS (Other)
  Interventions: Device: rTMS; Other: Genetic samples
- Depressive patients treated with SSRI (Other)
  Interventions: Drug: SSRI (SEROPLEX ou ZOLOFT); Other: Genetic samples
- Controls (Other)
  Interventions: Other: Genetic samples

INTERVENTIONS:
Device: rTMS
  Arms: Depressive patients treated with rTMS
Drug: SSRI (SEROPLEX ou ZOLOFT)
  Arms: Depressive patients treated with SSRI
Other: Genetic samples

SUMMARY:
Low frequency rTMS (repetitive Transcranial Magnetic Stimulation) for the treatment of patients with depression, is responsible for a decrease in the expression of the C-FOS and DUSP1 genes in peripheral blood leukocytes. The decrease in C-FOS expression could be explained by the inhibiting effect of low-frequency rTMS (in contrast, high-frequency rTMS causes activation of the cerebral cortex) [Rossi, 2009]. This genetic effect could correlate with the antidepressant effect [Hausmann, 2000].

According to this hypothesis, the genetic effect related to medical antidepressant treatments deserves to be studied because we could observe:

* either a decrease in the expression of the C-FOS and DUSP1 genes related to the antidepressant effect of the medical antidepressant treatment,
* or an increase in the expression of the C-FOS and DUSP1 genes related to cerebral activation due to the medical antidepressant treatment.

In summary, we wish to determine the validity of this hypothesis by comparing the genetic effect of rTMS with that of medical antidepressants to know if:

* this genetic effect is specific to rTMS or common rTMS and medical antidepressants
* this effect correlates with the clinical improvement induced by rTMS and by medical antidepressants
* this early modification in the C-FOS and DUSP1 genes may be predictor of the therapeutic response to rTMS and antidepressants (early decrease in gene expression)
* the absence of any decrease or increase in C-FOS and /or DUSP1 expression is a predictor of therapeutic resistance to rTMS and/or medical antidepressants.

ELIGIBILITY:
Inclusion Criteria:

Depressive patients to be treated with rTMS or SSRI:

* who have provided written informed consent
* who are covered by the national health insurance scheme
* who suffer from characterized depression (DSM-IV criteria) that is considered severe (Hamilton-17 item scale ≥ 19)
* who are aged 18-65 years,
* male or female
* who have presented at least one failed treatment with medical antidepressants prescribed at an effective dosage for a duration of at least 6 weeks.

Controls:

* Patients who have provided written informed consent
* who are covered by the national health insurance scheme
* aged between 18 and 65 years
* and either male or female

Exclusion Criteria:

Depressive patients destined to benefit from treatment with rTMS or SSRI:

* Type I or II bipolar disorders
* Depression with characteristics of psychosis
* Schizophrenia
* Abuse of alcohol and/or illegal psycho-active substances.
* Dependence on alcohol and/or an illegal psycho-active substance.
* Patients unable to provide consent to the protocol because of their mental disorders cannot be included in this study: patients with enforced psychiatric care (SDT, SDRE) or under ward of court.
* Contra-indication for rTMS; personal history of convulsions, pacemaker, neurosurgical clips, carotid or aortic clips, cardiac valves, audition prostheses, ventricular derivation valve, sutures with metallic thread or staples, foreign bodies in the eye, shrapnel, protheses or cephalic ferromagnetic implants, metal workers.
* Contra-indication for cerebral MRI
* Resistance to escitalopram or sertraline (prescription of escitalopram at 20 mg/d or sertraline at 50 mg/d for at least 6 weeks for the last episode)
* Contra-indication

  * for escitalopram : Hypersensitivity to escitalopram or one of the excipients. non-selective and irreversible monoamine oxidase (IMAO) inhibitors, because of the risk of serotoninergic syndrome with agitation, trembling, hyperthermia. reversible MAO-A inhibitors (e.g.: moclobemide) or a non-selective reversible MAO inhibitor (linezolid), given the risk of a serotoninergic syndrome
  * and to sertraline: Hypersensitivity to one of the components, Hypersensitivity to soja, Hypersensitivity to arachides, Treatment with IMAO
* Current pregnancy or breast-feeding: an assay for urinary beta-HCG will be done before inclusion in the protocol for women of child-bearing age.
* Contra-indication for escitalopram:

  * Hypersensitivity to escitalopram or to one of the excipients. No-selective, irreversible monoamine oxidase (IMAO), because of the risk of serotoninergic syndrome with agitation, trembling and hyperthermia.
  * Reversible MAO-A inhibitors (e.g.: moclobemide) or non-selective reversible MAO inhibitors (linezolid), because of the risk of serotoninergic syndrome.
  * Patients presenting an acquired or congenital prolonged QT interval and patients on treatments known to prolong or suspected of prolonging the QT interval (list of treatments on azcert.org).
* Contra-indication to sertraline:

  * Hypersensitivity to one of the components, Hypersensitivity to soja, Hypersensitivity to arachides, Treatment with IMAO. Patients treated with pimozide.

Controls:

* Any current psychiatric disease or a history of psychiatric disease (defined by DSM-IV-TR criteria)
* Current addiction (except for occasional smoking) or a history of addiction (defined by DSM-IV-TR criteria)
* Any progressive somatic disease (cardiac, hepatic, renal, pulmonary…)
* Any pharmacological treatment with the exception of combined oral contraceptive pills
* Current pregnancy or breast-feeding: urinary beta-HCG will be assayed before inclusion in the protocol in women of child-bearing age.
* Personnel employed in the psychiatry and addictology department of Dijon CHU

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-11-25 (Actual); Primary Completion 2018-06-05 (Actual)

PRIMARY OUTCOMES:
Leukocyte expression of the C-FOS and DUSP1 genes | At 2, 4 and 8 weeks of treatment with rTMS or an SSRI antidepressant

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Dijon, Dijon, France